CLINICAL TRIAL: NCT03354234
Title: Evaluation of a Prototype System for Generating Conditions of Orthostatic Hypotension and Blood Pooling in the Lower Body
Brief Title: Evaluation of the ORTHO-LBNP System
Acronym: ORTHO-LBNP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Military Institute of Aviation Medicine (Other Government)
Collaborators: Institute of Medical Technology and Equipment (Unknown); Nalecz Institute of Biocybernetics and Biomedical Engineering, Polish Academy of Sciences (Other); Polish Air Force Academy (Unknown); ETC-PZL Aerospace Industries Sp. z o.o. (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ORTHO-LBNP_01/2017
Record Dates: First submitted 2017-11-10; First posted 2017-11-27 (Actual); Last update posted 2018-05-18 (Actual); Status verified 2018-05

CONDITIONS: Orthostatic Hypotension; Ischemia; Hypoxia
Keywords: Gz accelerations; Head up tilt (HUT) test; Lower body negative pressure (LBNP) method; Physiological parameters; Variable gravitational stimuli
MeSH Terms: conditions — Hypotension, Orthostatic; Ischemia; Hypoxia | interventions — Lower Body Negative Pressure; Head-Down Tilt; Tilt-Table Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stimuli of slowly increasing intensities (Experimental): 1. 300-s check before the stimuli
  2. LBNP is applied stepwise with 11.1 mmHg/15 s decrement to -100 mmHg, and then this value is sustained for 120 s
  3. 180-second phase of rest between stimuli
  4. 75°-HUT (5°/s) for 120 s after a 15-s reversing of the gravity vector (-30°)
  5. 180-second phase of rest between stimuli
  6. 75°-HUT (5°/s) accompanied by an exposure to an LBNP of -60 mmHg increased linearly by -4 mmHg/s, and then this value is sustained for 120 s during HUT
  7. 120-s check after the stimuli
  Interventions: Other: Head up tilt (HUT); Other: Lower body negative pressure (LBNP); Other: Head down tilt (HDT); Device: Tilt table; Device: LBNP chamber
- Stimuli of rapidly increasing intensities (Experimental): 1. 120-s check before the stimuli
  2. 75°-HUT (45°/s) for 60 s after a 3-s reversing of the gravity vector (-30°)
  3. 180-second phase of rest between stimuli
  4. LBNP decreases linearly by -20 mmHg/s to -100 mmHg, and then this value is sustained for 60 s.
  5. 180 second phase of rest between stimuli
  6. push-pull, i.e., 3 x 75°-HUT (45°/s) preceded by -30°-HDT (45°/s) and accompanied by an exposure to an LBNP of -60 mmHg decreased linearly by -20 mmHg/s, and then this value is sustained for 30 s during HUT
  7. 120-s check after the stimuli
  Interventions: Other: Head up tilt (HUT); Other: Lower body negative pressure (LBNP); Other: Head down tilt (HDT); Device: Tilt table; Device: LBNP chamber

INTERVENTIONS:
Other: Head up tilt (HUT) — Model of -Gz: HUT up to 75 degrees (maximum)
Other: Lower body negative pressure (LBNP) — Model of -Gz: LBNP down to -100 mmHg (maximum)
Other: Head down tilt (HDT) — Model of +Gz: HDT down to -30 degrees (maximum)
Device: Tilt table — Range of tilt angles: -45° to +80°, rate of tilt changes: up to 45°/s
Device: LBNP chamber — Range of generated underpressure: 0 to -100 mmHg, rate of underpressure changes: up to 20 mmHg/s

SUMMARY:
The pilot study aims to evaluate a prototype system that enables military pilots to train under conditions of orthostatic hypotension and ischemic hypoxia. Both of these phenomena are experienced by aircraft crews of mainly highly maneuverable aircraft, and their syndromes include loss of color vision, loss of peripheral vision, blackout and finally G-induced loss of consciousness (G-LOC). A motorized tilt table to generate orthostatic (ORTHO) stress combined with an automatically controlled lower body negative pressure (LBNP) chamber to extort pooling of blood in the lower extremities has been developed in order to obtain new knowledge on counteracting the above-mentioned effects and minimizing the risk of their occurrence. This will help optimize the selection procedures of candidates with the best physiological predispositions to work as military pilots. The system is equipped with modules for monitoring biomedical parameters of a subject, including cerebral oxygenation, which ensures their safety and provides a source of data for performing advanced analyses. The ORTHO-LBNP system has been subjected to comprehensive laboratory tests and after a successful testing is ready for a pilot study involving pilots and/or cadets of the Polish Air Force Academy (PAFA). It is anticipated that new indicators will be proposed to enable an objective assessment of the predispositions to pursue a military pilot career. The prototype system can be easily adaptable to the needs of clinical and sports medicine as well as rehabilitation.

DETAILED DESCRIPTION:
The pilot study consists of two research scenarios, in which two different sequences of the interventions taking the form of the pre-programmed tilt and LBNP profiles are to be investigated.

1. Scenario I is designed to initially verify the potential impact of the prototype system on the human body. For this purpose, only basic tilt and LBNP stimuli of relatively slowly increasing intensities will be used, and the group of subjects will include only subjects with flight experience. Up to 20 PAFA cadets shortly before graduation, including women and men, will be involved in the pilot study (experimental arm 1). The subjects will be healthy, aged between 20 and 30 years old. Scenario I will take almost 24 min.
2. Scenario II is to compare subjects with and without flight experience using rapid tilt and LBNP stimuli as well as a push-pull stimulus. Up to 30 subjects including up to 15 pilots, i.e., flight school adepts shortly after graduation and/or PAFA cadets shortly before graduation, and up to 15 students of the Aviation High School in Dęblin, Poland, including women and men will be involved in the study (experimental arm 2). The subjects will be healthy, aged between 18 and 30 years old. The students of the Aviation High School will participate in the study as a reference group, without flight experience. Scenario II will take 16 min.

The pilot study will be carried out in an isolated room in the presence of a physician (physiologist), a paramedic and an ORTHO-LBNP system operator. The paramedic will prepare the subject for the study by placing on his/her body electrodes and measuring sensors that will be removed after completion of the study. The subject will be asked to close his/her eyes during the tests and to place his/her hands on the rest. In order to cause the least disturbance, no conversation will be held with the subject. Only if disturbing symptoms will occur, will the subject immediately report this to the personnel. The physician will systematically be observing the subject's cardiogram, his/her HR, continuous non-invasive arterial pressure (CNAP) wave, and systolic and diastolic blood pressure (SBP and DBP, respectively) in comparison with the changing tilt of the table and negative pressure in the chamber. Any time, at the request of the subject or on the instruction of the physician, the operator will interrupt the tests. The tilt table then will return to the Trendelenburg position if interruption occur during HUT and/or LBNP stimuli, or horizontal position if interruption occur during HDT stimulus. At the same time atmospheric pressure will be resumed in the chamber.

ELIGIBILITY:
Inclusion Criteria:

* Pilots or cadets with flight experience
* Candidates for pilots without flight experience
* None alcohol 24 hours prior to the study
* Written informed consent

Exclusion Criteria:

* Subjects with cardiovascular disorders

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2017-01-02 (Actual); Primary Completion 2018-02-17 (Actual); Study Completion 2018-02-17 (Actual)

PRIMARY OUTCOMES:
HR | 24 minutes (scenario I)
  Heart rate in beats per minute
IBI | 24 minutes (scenario I)
  Inter-beat interval in seconds
SBP | 24 minutes (scenario I)
  Systolic blood pressure in millimeters of mercury
DBP | 24 minutes (scenario I)
  Diastolic blood pressure in millimeters of mercury
MAP | 24 minutes (scenario I)
  Mean arterial pressure in millimeters of mercury
SV | 24 minutes (scenario I)
  Stroke volume in milliliters
CO | 24 minutes (scenario I)
  Cardiac output in liters per minute
LVET | 24 minutes (scenario I)
  Left ventricular ejection time in milliseconds
RPP | 24 minutes (scenario I)
  Rate pressure product in millimeters of mercury
TPR | 24 minutes (scenario I)
  Total peripheral resistance in medical units

SECONDARY OUTCOMES:
Z0_T | 16 minutes (scenario II)
  Base transthoracic impedance in ohms
dZ/dt_T | 16 minutes (scenario II)
  First derivative of transthoracic impedance in ohms per second
Z0_H | 16 minutes (scenario II)
  Base transcephalic impedance in ohms
dZ/dt_H | 16 minutes (scenario II)
  First derivative of transcephalic impedance in ohms per second
ΔC_HbO2 | 16 minutes (scenario II)
  Changes in oxygenated hemoglobin in micromolars
ΔC_Hb | 16 minutes (scenario II)
  Changes in deoxygenated hemoglobin in micromolars
ΔC_tot | 16 minutes (scenario II)
  Changes in total hemoglobin in micromolars

CONTACTS AND LOCATIONS:
Overall Officials: Łukasz Dziuda, DSc, PhD, Principal Investigator — Military Institute of Aviation Medicine
Locations (1):
- Military Institute of Aviation Medicine, Warsaw, Poland

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-11-10): https://cdn.clinicaltrials.gov/large-docs/34/NCT03354234/Prot_SAP_ICF_000.pdf